CLINICAL TRIAL: NCT06894264
Title: Emotion Processing and Regulation in People with Intellectual Disability
Acronym: EPRID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Rück, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPRID
Record Dates: First submitted 2025-02-10; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Intellectual Disabilities (F70-F79); Autism Spectrum Disorder
Keywords: Emotion regulation; Psychological experiment; Psychotherapy
MeSH Terms: conditions — Intellectual Disability; Autism Spectrum Disorder; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Emotion regulation (Experimental): The CBT for emotion regulation is an adapted version of the DBT skills Manual by Linehan for patients with ID.
  Interventions: Behavioral: Emotion regulation

INTERVENTIONS:
Behavioral: Emotion regulation — The intervention is an adapted version of skills training that stems from DBT. The text has been simplified, and illustrations have been added to facilitate learning. In addition, metaphors have been removed, making it more user-friendly for the targeted populations. It consists of 12 modules that are delivered during 12 weeks, one module per week. A licensed psychologist are responsible for each individual treatment. Care givers or relatives are encouraged to participate and help the study participant to complete their homework assignments.

SUMMARY:
BACKGROUND

Intellectual disability (ID) is neurodevelopmental disorder with social impairments, in areas such as interpersonal communication skills and emotion regulation. This overlaps with disabilities associated with autism spectrum disorder (ASD). Differences in emotion processing, specifically emotion recognition, reappraisal, and reinforcement learning, has not been compared between patients with ID and ASD. Despite difficulties in emotion regulation among patients with ID, there is a lack of adapted psychotherapy for this patient group.

AIMS

* To examine differences in emotion processing in individuals with intellectual disability (ID) compared to individuals with autism spectrum disorder (ASD) and typically developed individuals.
* To evaluate the feasibility and effectiveness of an adapted psychotherapeutic intervention to improve emotion regulation in individuals with ID.

Data and method

The first research question is addressed through a cross-sectional study involving 160 participants: 40 individuals with ID, 40 individuals with ASD, and 80 typically developed controls. Participants will undergo psychological experiments where the investigator simultaneously measure eye movement and pupil dilation using an eye-tracker. To investigate different aspects of social cognition, the investigator will use three psychological experiments: emotion recognition, emotion reappraisal, and reinforced learning in a social context. Differences in social cognition are subsequently used in predictive models to predict the group affiliation of study participants.

To evaluate the effectiveness and feasibility of an adapted emotion regulation treatment, the 40 study participants with ID will undergo a manual-based psychotherapy. The treatment, adapted from skills training in dialectical behavior therapy, consists of 12 individual sessions over 12 weeks. The treatment includes four main modules: mindfulness skills, relationships, emotion regulation, and emotional resilience. Outcome measures are administered at baseline, post-treatment, and at a 6-month follow-up.

SOCIETAL RELENVANCE

This research addresses a significant knowledge gap in social cognition and mental health in individuals with ID. The results may lead to a better understanding of differences in social cognition compared to individuals with ASD, and effective, targeted interventions for emotion regulation in individuals with ID. In the long run, the treatment could help reduce off-label prescription of antipsychotics to manage behavioral deviations in individuals with ID, as challenging behaviors often stem from difficulties with emotion regulation.

PROJECT REALISATION

The research group consists of an interdisciplinary composition of experts in neuropsychology, experimental psychology, and implementation of psychotherapeutic research. The project has obtained ethical approval and follows the principles of open science, with pre-registration of study protocols.

DETAILED DESCRIPTION:
BACKGROUND

Individuals with intellectual disability (ID) experience significant difficulties in interpreting, controlling, and expressing emotions. These deficits in emotion processing contribute to challenging behaviors, manifesting as aggressive outbursts, self-injurious behaviors, or withdrawal. The ability to understand and regulate emotions plays a vital role in daily functioning and social interactions. Impairment in emotion regulation also leads to increased stress, anxiety, and mood disorders, further exacerbating behavioral issues and negatively impacting the overall quality of life for individuals with ID.

Traditional cognitive tests (e.g., Wechsler Adult Intelligence Scale, WAIS) are reliable in measuring certain cognitive abilities but fall short in assessing emotional processes and social learning under uncertainty. New, objective measurement tools grounded in cognitive and neuroscience theories, would enhance our understanding of the challenges that patients with ID face in a social context.

Study has shown that Patients with ID have greater difficulty recognizing emotions compared to typically developing peers. Patients with ASD share the same functional impairment. However, the underlying mechanisms for these difficulties may differ between the two groups. For individuals with ASD, reduced fixation on the eye region has been proposed as a contributing factor to their emotion recognition difficulties, while the difficulties for individuals with ID may be due to more complex cognitive factors beyond simply reduced eye fixation.

Emotional reappraisal is a cognitive strategy used to regulate emotions by reinterpreting the meaning of emotional stimuli. It is crucial for effective emotion regulation as it allows individuals to change their emotional responses by altering their perspective on the emotional situations. For individuals with ID, the cognitive demands of reappraisal may be challenging due to limitations in executive functioning and abstract thinking, whereas for ASD, difficulties in theory of mind could impede the ability to reframe emotional situations effectively. Elucidating the exact impairment in emotion reappraisal could therefore impact assessment tools, treatment strategy and response to emotion regulation therapy.

Research in psychology and neuroscience has identified feedback learning as a crucial form of learning in humans. Typically, people adhere to a simple, yet powerful and flexible strategy called reinforcement learning (RL). Central to RL is that learning is driven by a mismatch between the initial belief about the outcome and the actual outcome. This mismatch is known as a prediction error. Differences in how prediction errors are computed and used for learning could be a distinct feature in cognitive processing between patients with ID and ASD. Moreover, understanding prediction errors and reinforcement learning mechanisms from a social context may be crucial in explaining how individuals assimilate and respond to clinical interventions, potentially offering insights into treatment efficacy and personalized therapeutic approaches.

Prevalence of challenging behavior in individuals with ID is between 10-15% and a common reason for refferal to psychiatry. 65% of youths with intellectual and developmental disabilities who were referred to a mental health service were prescribed antipsychotics. However, randomized controlled trials have not demonstrated consistent efficacy for this approach (SMD=-0.85; 95% CI=-1.69 to -0.01; p=0.05). Despite the clear need for psychological interventions to adress this issue, there is a striking disparity in the availability and application of psychotherapy for individuals with ID compared to the general population. This gap in treatment options highlights the necessity for targeted interventions that enhance emotion regulation and social functioning in this population. Among the various therapeutic approaches, skills-based training programs rooted in Dialectical Behavior Therapy (DBT) have shown promise in addressing these challenges. DBT focuses on teaching skills in mindfulness, distress tolerance, emotion regulation, and interpersonal effectiveness. In a pilot study with six participants, this form of treatment led to decreased challenging behaviors, improved global functioning, and reduced hospital admissions, suggesting potential efficacy of this treatment approach in a Swedish context. However, existing studies have typically involved small numbers of participants, highlighting the need for further research to elucidate the efficacy and feasibility of emotion regulation therapy for patients with ID. Despite these limitations, emotion regulation therapy represents a promising avenue for improving the quality of life and social functioning of individuals with intellectual disabilities.

Preliminary results

Associate Professor Kleberg's research group has extensive experience conducting eye-tracking studies in individuals with Autism Spectrum Disorder (ASD) and rare genetic syndromes across varying cognitive abilities. Their previous research has revealed distinct eye-movement patterns and pupillary responses in individuals with rare genetic syndromes, such as Williams syndrome and Turner syndrome, which differ from those observed in individuals with ASD during psychological experiments. This line of research is crucial for understanding the unique cognitive and social profiles associated with different neurodevelopmental conditions.

A population-based longitudinal study by dr. Hirvikoski uncovered excess premature death among people with ID. The increased risk for causes of death were potentially amendable to health care, including cause-specific mortality in circulatory system and neoplasm. Challenging behaviors, including aggression, destructive behavior, and self-harm, occur in an estimated 10-15% of patients with ID. Second-generation antipsychotics (SGAs) are now widely prescribed off-label to manage these behaviors. However, the long-term neurologic, metabolic, and hormonal effects of SGAs in this population remain largely unknown.

A pilot study by Nylander et al., suggest that a modified version of dialectic behavioral therapy is effective in reducing self-harm and can reduce the number of hospital admissions on an individual level. However, a larger cohort study assessing the ability for emotion regulation to reduce self-harm is warranted. In addition this manual has been shortened to 12 sessions and involve relatives or carers that can support the patient during and after the therapy. This manual has been tested clinically at the neuropsychiatric outpatient clinic. Seven patients with neuropsychiatric disabilities show improvement in emotion regulation measured with DERS-SF and report that they were mostly satisfied according to the CSQ-8 questionnaire.

METHODS

Study design

The first part of the study (aim 1) has a cross-sectional design while the second part (aim 2) is an interventional trial.

Participants

Inclusion criteria:

ID Group: 40 individuals with mild ID (DSM-5 criteria, IQ 52-70) ASD Group: 40 individuals with ASD (DSM-5 criteria, IQ 85-115) TD Group: 80 individuals without neurodevelopmental disorders (IQ 85-115) All study participants are adults between the ages of 18-45, and can read and communicate in Swedish. The control group are matched by sex and age ± 5 years.

Exclusion criteria: Presence of severe sensory impairments (e.g., blindness, deafness); current psychosis or affective disorder; significant neurologic disorders (e.g., epilepsy) or degenerative disorder (e.g.. dementia, Parkinson's disease); diagnosis of ADHD; ongoing substance abuse, specific medication that enhance cognitive performance (central stimulants) or psychotropic medication that could affect task performance (anti-epileptic medication), emotion regulation therapy or corresponding psychotherapy during the last 12 months.

Procedure

Informed written consent will be obtained from all participants prior to inclusion. During the pre-assessment phase all study participants will undergo the following assessments (Mini-International Neuropsychiatric interview (M.I.N.I.), Wechsler Adult Intelligence Scale (WAIS-IV), Social Responsiveness scale (SRS-2), The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) Interview Form).

All outcome measures from the emotion regulation therapy will be administered at baseline, post-treatment (primary endpoint), and at 6-month follow-up (except for client satisfaction questionnaire and negative effects questionnaire):

Difficulties in emotion regulation scale (DERS-SF), The Behavior Problems Inventory (BPI-01), World Health Organization Disability Assessment Schedule 2.0, The Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) Scales, Client Satisfaction Questionnaire (CSQ-8), Negative effects questionnaire (NEQ).

Testing protocol for psychological experiments with eye-tracking

Eye tracking technology offers a non-invasive and cost-effective method for studying cognitive processes and behavioral patterns in individuals with developmental disorders.

Emotion recognition task:

Design. The emotional recognition task will consist of a series of trials, each presenting a facial expression representing one of the basic emotions: happiness, sadness, anger, fear, surprise, and disgust. The face for each trial is chosen randomly. Each trial will begin with a fixation cross displayed at the center of the screen for 500 ms, followed by the presentation of a face, on either the left or right side, that changes from neutral to the emotion that the test subject is asked to identify.

Objective. Participants are asked to answer if the statement is correct by giving thumbs up for correct statement and thumbs down for incorrect statement.

Data collection. Reaction time (time taken to select an answer), and accuracy (correct identification of the emotion) will be recorded. Eye-tracking data consists of two parameters. Orientation toward eyes measured by the saccade gaze motion, and gaze path divided into areas of interest. Faces are divided into four regions of interest (whole face, eyes, nose and mouth).

Emotion reappraisal task:

Design. This task consists of two conditions: view and reappraise. During the view phase, participants are given the instruction to watch an image before the image is presented. Afterwards the participants are asked to rate how emotionally negative the image was on a Likert scale of 1-8. During the reappraisal phase, participants are given the instruction to reappraise before an image is presented. Participants are asked to state the cognitive reappraisal aloud. Afterwards the participants are asked to rate how emotionally negative the image was again on the Likert scale.

Objective. Participants are asked to watch the image in the view condition and instructed to change their emotional experience through cognitive reappraisal during the reappraisal condition. Expressing positive outcomes or alternative meanings that are less negative reflect their ability for reappraisal, and the decrease in negative emotion reflect their reappraisal efficacy.

Data collection. Baseline reactivity to images, reappraisal ability and efficacy will be registered. The reappraisal statements will be analyzed by a researcher blind to the study hypothesis. Pupil dilatation will be recorded for each trial.

Social reinforcement learning task:

Design. Two shapes with different orientations are presented for each trial. At the beginning of the trial a hidden rule for correct answer is established. Depending on how the test subject answers, a face depicting a positive or negative feedback is provided. When a certain number of correct answers are provided which reflect an understanding of the underlaying rule, the rule switches. The task is to identify the new rule.

Objective. Participants are asked to provide the correct answer and through social reinforced learning identify the underlaying rule.

Data collection. Reaction time (time to response) and accuracy (correct answers) will be recorded. Eye-tracking data consists of two main parameters. Pupilar dilatation and gaze path (length) will be measured during each trial.

Emotion regulation therapy

The psychotherapy for emotion regulation is an adapted version of the DBT skills Manual by Linehan for patients with ID (13). The text has been simplified, and illustrations have been added to facilitate learning. In addition, metaphors have been removed, making it more user-friendly for the targeted populations.

The adapted treatment consists of four modules: skills in mindfulness, skills in relationship, skills in regulating emotions, skills in emotional resilience. The treatment consists of twelve sessions given over twelve weeks. The treatment will be provided individually by a licensed psychologist. Health care provider or relatives who live with the participant are invited to facilitate learning and practicing the skills as well as aid them in responding to questionnaires.

Feasibility will be assessed according to the RE-AIM framework (reach, effectiveness, adoption, implementation, maintenance) (16). Reach will be measured by looking at the percentage eligible/excluded, reasons for refusal or exclusion. Effectiveness will be measured using symptom reductions on the primary outcome measures (DERS-SF and WHODAS 2.0). Adoption will be assessed by looking at short-term attrition during the treatment, self-reported time spent on assignments, and the Client Satisfaction Questionnaire (CSQ-8) at post-treatment. Adverse events data will be collected post-treatment and at the 6-month follow-up where the patients will rate a list of common adverse events using the negative effects questionnaire (NEQ). Implementation will be assessed by looking at the number of additional telephone calls made by therapists.

Fidelity in the treatment is ensured by thorough training and continuous supervision between sessions. After each session, the therapist must fill in a "Fidelity checklist" that outlines the specific elements that therapists need to cover in each session. Evaluation of treatment outcomes at post-treatment is performed by an independent researcher.

Data analysis plan

The investigator will employ machine learning algorithms using tidymodels to build predictive models, evaluating their performance through internal validation and area under the curve (AUC) metrics (Aim 1A). To evaluate whether emotion regulation therapy improves emotion processing in patients with ID (Aim 1B), the investigator will employ a repeated measures ANOVA or mixed-effects models to compare pre- and post-treatment performance on emotion recognition tasks, reappraisal tasks, and eye-tracking metrics. Effect sizes will be calculated using partial eta-squared (η²) for ANOVA or marginal R² for mixed-effects models.

To evaluate the efficacy of emotion regulation therapy for ID patients, the investigator will use mixed-effects linear regression models to compare pre- and post-treatment scores on DERS-SF and WHODAS 2.0, calculating within-group effect sizes using Cohen's d (Aim 2A). Feasibility will be analyzed according to the RE-AIM framework, examining metrics such as eligibility/exclusion percentages, attrition rates, time spent on assignments, CSQ-8 scores, adverse events, and additional support required during treatment (Aim 2B). Throughout the analysis, the investigator will ensure appropriate data transformations (e.g., log-transformation for reaction times) and alternative non-parametric tests when normality assumptions are not met.

Power calculation

Previous studies have demonstrated the effectiveness of cognitive behavioural therapy (CBT) and DBT-informed interventions for improving emotional regulation in individuals with ID, showing medium effect sizes (Cohen's d ranging from 0.3-0.6). Assuming an effect size of 0.5 and a standard deviation of 1 (0.8-1.1) for standardised effect size, an alpha level of 0.05, and 80% power, a conservative estimate would suggest that a sample size of approximately 30-35 participants is required to detect a significant improvement in DERS-SF. The investigator plan to recruit more participants than required for the primary analysis to account for missing or incomplete data and to ensure that the study maintains statistical power. This approach will also enable robust subgroup analyses and enhance the overall generalizability of the results.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with mild ID based on DSM-5 criteria, corresponding to a general IQ between 52-70.
* Can read and communicate in Swedish.

Exclusion Criteria:

* Presence of severe sensory impairments (e.g., blindness, deafness)
* Current psychosis or affective disorder; significant neurologic disorders (e.g., epilepsy) or degenerative disorder (e.g.., dementia, Parkinson's disease) - Diagnosis of ADHD
* Ongoing substance abuse
* Specific medication that enhance cognitive performance (central stimulants) or psychotropic medication that could affect task performance (anti-epileptic medication)
* Emotion regulation therapy or corresponding psychotherapy last 12 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Difficulties in emotion regulation scale (DERS-SF) | From enrollment to the end of treatment at 12 weeks
  DERS-SF is a self-report questionnaire that assesses individuals' difficulties in emotion regulation. It consists of 18 questions, rated on a Likert scale of 1-5, and takes 10 minutes to complete.
  Total point: 18-90 Higher scores = greater emotion dysregulation

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 | From enrollment to the end of treatment at 12 weeks
  the interview-administered version is a comprehensive tool designed to assess disability and functioning across multiple domains in adults aged 18 and older. WHODAS 2.0 evaluates six key areas of functioning: cognition, mobility, self-care, getting alone, life activities, and participation. The interview-administered version is conducted by a trained interviewer who asks questions and records the respondent's answers. This format allows for clarification and ensures all items are addressed. It takes 20-30 minutes to complete.
  Total point: Varies by version (e.g., 12- or 36-item), but scores are converted to a 0-100 metric Higher scores = greater disability
The Clinical Global Impression - Severity scale (CGI-S) | From enrollment to the end of treatment at 12 weeks
  CGI-S will be used to assess overall clinical severity by the clinican. Total points: 1-7 Higher scores = more severe symptoms
Clinical Global Impression - Improvement scale (CGI-I) | From enrollment to the end of treatment at 12 weeks
  will be used to assess treatment response by the clinician. Total points: 1-7 Higher scores = worsening symptoms or lack of improvement
Client Satisfaction Questionnaire (CSQ-8) | From enrollment to the end of treatment at 12 weeks
  CSQ-8 evaluates client satisfaction with the intervention or treatment received. This self-report questionnaire takes approximately 5-10 minutes to complete and consists of 8 items rated on a Likert scale. It assesses various aspects of satisfaction, including the quality of service, helpfulness, and overall experience.
  Total points: 8-32 Higher scores = greater satisfaction (lower scores indicate dissatisfaction)
The Behavior Problems Inventory (BPI-01) | From enrollment to the end of treatment at 12 weeks
  The BPI-01 is an informant-based behavioral assessment tool used to evaluate maladaptive behaviors in individuals with intellectual and developmental disabilities, including autism spectrum disorders. The BPI-01 measures in detail the frequency and severity of three common types of problematic behaviors: self-injurious behavior, stereotyped behavior, and aggressive/destructive behavior. The instrument consists of 52 questions answered by an informant who knows the person well, typically a caregiver or family member. The BPI-01 takes approximately 15 minutes to complete and provides a comprehensive picture of behavioral problems in the individual.
  Self-Injurious Behavior:
  Frequency: 0-56 (14 items × 0-4) Severity: 14-42 (14 items × 1-3)
  Stereotyped Behavior:
  Frequency: 0-96 (24 items × 0-4) Severity: 24-72 (24 items × 1-3)
  Aggressive/Destructive Behavior:
  Frequency: 0-44 (11 items × 0-4) Severity: 11-33 (11 items × 1-3)
  Higher scores = more frequent/severe problematic behaviors
Negative effects questionnaire (NEQ) | From enrollment to the end of treatment at 12 weeks
  NEQ is a self-report instrument designed to assess adverse events associated with psychological treatments. It consists of 32-item and an open-ended question in the end. Participants rate items on a five-point Likert scale, with the questionnaire taking approximately 10-15 minutes to complete.
  Total points: 20-80 Higher scores = greater negative treatment effects

IPD SHARING:
Plan to Share IPD: No
To avoid identification of individual study participants

REFERENCES:
- [Background] Linehan MM, Wilks CR. The Course and Evolution of Dialectical Behavior Therapy. Am J Psychother. 2015;69(2):97-110. doi: 10.1176/appi.psychotherapy.2015.69.2.97. PMID 26160617
- [Background] Jahoda A, Dagnan D, Hastings R, Gillooly A, Miller J, Baines S, Hatton C. Adapting psychological interventions for people with severe and profound intellectual disabilities: A behavioural activation exemplar. J Appl Res Intellect Disabil. 2024 Mar;37(2):e13199. doi: 10.1111/jar.13199. PMID 38361369
- [Background] Campos-Jara R, Martinez-Salazar C, Campos-Jara C, Fernandez JM, Martinez-Garcia D, Contreras-Osorio F. Pharmacological treatment for challenging behavior in adults with intellectual disability: Systematic review and meta-analysis. Span J Psychiatry Ment Health. 2024 Oct-Dec;17(4):231-238. doi: 10.1016/j.rpsm.2023.01.003. Epub 2023 Jan 31. PMID 37839961
- [Background] Kleberg JL, Willfors C, Bjorlin Avdic H, Riby D, Galazka MA, Guath M, Nordgren A, Strannegard C. Social feedback enhances learning in Williams syndrome. Sci Rep. 2023 Jan 4;13(1):164. doi: 10.1038/s41598-022-26055-8. PMID 36599864
- [Background] Garrison J, Erdeniz B, Done J. Prediction error in reinforcement learning: a meta-analysis of neuroimaging studies. Neurosci Biobehav Rev. 2013 Aug;37(7):1297-310. doi: 10.1016/j.neubiorev.2013.03.023. Epub 2013 Apr 6. PMID 23567522
- [Background] Subramanian A, Chitlangia S, Baths V. Reinforcement learning and its connections with neuroscience and psychology. Neural Netw. 2022 Jan;145:271-287. doi: 10.1016/j.neunet.2021.10.003. Epub 2021 Oct 22. PMID 34781215
- [Background] Littlewood M, Dagnan D, Rodgers J. Exploring the emotion regulation strategies used by adults with intellectual disabilities. Int J Dev Disabil. 2018 Jun 8;64(3):204-211. doi: 10.1080/20473869.2018.1466510. PMID 34141307
- [Background] Samson AC, Sokhn N, Van Herwegen J, Dukes D. An exploratory study on emotion regulation strategy use in individuals with Williams syndrome, autism spectrum disorder and intellectual disability. Front Psychiatry. 2022 Nov 23;13:940872. doi: 10.3389/fpsyt.2022.940872. eCollection 2022. PMID 36506439
- [Background] Jenner LA, Farran EK, Welham A, Jones C, Moss J. The use of eye-tracking technology as a tool to evaluate social cognition in people with an intellectual disability: a systematic review and meta-analysis. J Neurodev Disord. 2023 Dec 4;15(1):42. doi: 10.1186/s11689-023-09506-9. PMID 38044457
- [Background] Scotland JL, McKenzie K, Cossar J, Murray A, Michie A. Recognition of facial expressions of emotion by adults with intellectual disability: Is there evidence for the emotion specificity hypothesis? Res Dev Disabil. 2016 Jan;48:69-78. doi: 10.1016/j.ridd.2015.10.018. Epub 2015 Nov 5. PMID 26546741
- [Background] Hermann H, Berndt N, Lytochkin A, Sappok T. Behavioural phenomena in persons with an intellectual developmental disorder according to the level of emotional development. J Intellect Disabil Res. 2022 May;66(5):483-498. doi: 10.1111/jir.12930. Epub 2022 Mar 31. PMID 35357054